CLINICAL TRIAL: NCT01188824
Title: The Safety and Efficacy of Cilostazol in Ischemic Stroke Patients With Peripheral Arterial Disease (SPAD Study)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Collaborators: National Taiwan University Hospital (Other); Shin Kong Wu Ho-Su Memorial Hospital (Other); Tri-Service General Hospital (Other); Far Eastern Memorial Hospital (Other); Changhua Christian Hospital (Other); Chi Mei Medical Hospital (Other); National Cheng-Kung University Hospital (Other); Kaohsiung Medical University Chung-Ho Memorial Hospital (Other); E-DA Hospital (Other); Mackay Memorial Hospital (Other); Cathay General Hospital (Other); En Chu Kong Hospital (Other); Kuang Tien General Hospital (Other); Chung Shan Medical University (Other); Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DMR99-IRB-137
Record Dates: First submitted 2010-08-23; First posted 2010-08-26 (Estimated); Last update posted 2013-10-07 (Estimated); Status verified 2013-07

CONDITIONS: Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke | interventions — Cilostazol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cilostazol (Active Comparator): Pletaal® (Cilostazol) 100 mg, bid p.o.
  Interventions: Drug: Cilostazol
- placebo (Placebo Comparator): Placebo
  1 tablet, bid p.o.
  Interventions: Other: placebo

INTERVENTIONS:
Drug: Cilostazol — 100 mg, bid p.o.
  Other Names: Pletaal®
  Arms: Cilostazol
Other: placebo — 1 tablet, bid
  Arms: placebo

SUMMARY:
The purpose of this study is to investigate the Safety and Efficacy of Cilostazol in slowing down the progression of peripheral arterial disease (PAD) in ischemic stroke patients with PAD in Taiwan.

DETAILED DESCRIPTION:
One thousand patients will be randomized to take cilostazol (500 patients) or placebo (500 patients) in parallel groups. Patients will be screened and evaluated on Visits 1 to assess their eligibility prior to randomization. The treatment period (Visit 1-6) will last 12 months and the patient will receive initial and follow-up evaluation (section 4.5) including history and physical examinations, and baseline and end of treatment ABI and carotid IMT assessments. Vascular events and death as well as adverse events including bleeding complications will also be recorded at intervals as detailed in section 4.5.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients, age ≧50 years; for female patients, postmenopausal (defined as at least 2 years without menses) has to be confirmed.
* Ischemic stroke or transient ischemic attack patients who have been taking aspirin 100 mg, QD
* Neurologically and clinically stable at inclusion
* PAD (i.e. ankle-brachial index or ABI <1.0)

Exclusion Criteria:

* Patients unable to give informed consent
* Patients with history of any type of hemorrhagic stroke (intracerebral hemorrhage,subarachnoid hemorrhage, or others)
* Modified Rankin Scale >4
* Patients with history of dementia requiring institutional care
* Known brain tumor
* Known anemia (defined as hemoglobin <10.0 g/dL)
* Known thrombocytopenia (defined as platelet count below 100,000/cm3)
* AST or ALT > 3 x Upper Normal Limit
* Calculated creatinine clearance < 30 ml/min according to the Copckroft formula)
* Known hemostasis or coagulation disorder
* Congestive heart failure, defined as a previous definitive diagnosis, or present symptoms of at least Category II of the NYHA classification system for CHF
* Revascularization of the lower limb arteries including bypass surgery, endovascular procedures
* Symptomatic PAD requiring treatment with cilostazol
* Known stenosis of the upper limb arteries that may affect the documentation of ABI
* Patients with known hypersensitivity to cilostazol

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 801 (Actual)
Dates: Start 2010-09; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
The primary endpoint for this study is slowdown of PAD progression based on ABI. | 2 years

SECONDARY OUTCOMES:
Carotid intima-media thickness | 2 years
  1. Carotid intima-media thickness.
  2. Vascular events, including recurrent stroke, myocardial infarction, unstable angina,other vascular events, and all death.
  3. Safety, including major bleeding events, hemorrhagic stroke, any death.

CONTACTS AND LOCATIONS:
Overall Officials: Chung Y. Hsu, MD. Ph.D., Principal Investigator — China Medical University Hospital